CLINICAL TRIAL: NCT06189430
Title: Effect of Vinyasa Yoga on Frailty and Anthropometric Measurements in Elderly Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Meltem Adaici, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 879
Record Dates: First submitted 2023-12-06; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Geriatrics; Yoga; Complementary Therapies; Nursing Caries
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Intervention Model Description: This study was planned as a randomized controlled, double-blind and experimental study to evaluate the effect of vinyasa yoga on frailty and anthropometric measurements in elderly individuals.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Research data were collected by one-on-one and face-to-face interviews using data collection tools and the statistician was blinded. Hrobjartsson et al. (2013) report that blinding the person performing the statistical analysis, which is frequently preferred in non-pharmaceutical research, has positive effects in terms of reducing bias in effect size estimates and is also useful if the measurements are subjective. It is emphasized that blinding those who measure subjective data, which can only be obtained from the individual and which generally constitute the main criteria of nursing studies, is a feasible and preferable method. For this reason, the data in our study was collected by another research assistant outside the study. For all tests performed, individuals were given nicknames and data entries were made.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Group (Experimental): Individuals in the yoga group of the study had 10 minutes of meditation, 10 minutes of warm-up, and 40 minutes of vinyasa yoga practice, 2 days a week face-to-face and 1 day online, for a total of 12 weeks.Yoga practice was standardized throughout the study to avoid the risk of intervention variability. The basic structure of each yoga session is meditation, breathing exercises (pranayama), and after a warm-up, yoga practice includes asanas (postures) for strength, balance and mobility, and finally ends with relaxation.
  Interventions: Other: Yoga
- Control Group (Active Comparator): In order to better understand the effectiveness of Vinyasa yoga, individuals in the control group will perform moderate-intensity standard exercise (50-70% MHR: maximum pulse rate) for the same duration and at the same hours.
  Interventions: Other: Standard exercise

INTERVENTIONS:
Other: Yoga — Yoga practice was standardized throughout the study to avoid the risk of intervention variability. The basic structure of each yoga session is meditation, breathing exercises (pranayama), and after a warm-up, yoga practice includes asanas (postures) for strength, balance and mobility, and finally ends with relaxation. The yoga intervention we recommend was created within the framework of the asanas that the elderly can do in the literature and by taking the expert opinion of a sports physician.
  Other Names: Vinyasa Yoga
  Arms: Yoga Group
Other: Standard exercise — It is a type of exercise similar in intensity to vinyasa yoga. (50-70% MHR: maximum pulse rate)
  Arms: Control Group

SUMMARY:
During the aging process, concrete changes such as loss of function in organs and systems resulting from biological, physiological and psychological negativities and difficulty in participating in daily life activities occur. Frailty, one of the geriatric syndromes, is a complex condition that increases vulnerability to stressors and causes a decrease in the physiological reserve necessary to maintain homeostasis in most organs. When examined pathophysiologically, it is thought that frailty is not only evaluated as physical, but psychological and social fragility may also contribute to this situation.

It is thought that physical activity that includes strength training to maintain or improve muscle mass throughout aging may reduce muscle loss, an important risk factor for frailty. To treat physical frailty, supervised exercise is recommended as an effective strategy. Yoga; It is a holistic practice that encourages healing through breathing, movement, strength, flexibility and achieving integrity of spirit, body and mind. Being a meditative practice distinguishes yoga from other typical forms of physical exercise, despite having similar metabolic intensity. Regular yoga has the potential to improve flexibility, balance and muscle strength in older individuals. It is also known that yoga improves cognitive function in the elderly, helps manage chronic conditions, reduces pain due to osteoarthritis, improves sleep, increases subjective well-being and health-related quality of life.

During the healthy aging process, people may need to be guided according to their individual and health characteristics. By supporting this situation with appropriate nursing care, losses can be reduced and optimum health can be maintained. One of the biggest advantages of yoga applied within the scope of nursing care is that the individual's progress is ensured in a controlled manner by preparing a flow in line with appropriate asana selections, taking into account the individual's health condition. Nursing, by its nature, requires a holistic approach to people. Similarly, the practice of yoga is considered a practice that integrates not only physical health but also the mind, body and soul.

This study was planned as a randomized controlled, double-blind and experimental study to evaluate the effect of vinyasa yoga on frailty and anthropometric measurements in elderly individuals.

DETAILED DESCRIPTION:
Epidemiological studies and evidence-based practices conducted with the increasing elderly population in the world suggest that active and healthy aging can be achieved by preventing age-related inadequacies and limitations due to changes in negative factors that occur with aging. Active aging is the process of enabling the individual to perform all his/her functions independently and maintaining and protecting his/her health in a physically, psychologically and socially safe environment. In addition, during this period, the person has the opportunity to improve himself while increasing his subjective well-being levels and related quality of life by focusing on his strengths rather than the losses he experiences due to old age.

To date, exercise remains the interventional modality that most consistently provides benefit in the treatment of frailty and its core components. Exercise has physiological effects on almost all organ systems, especially the musculoskeletal, endocrine and immune systems. It is known that supervised exercise programs in healthy and pre-frail elderly individuals have positive effects on their participation in daily life activities while reducing physical fragility. Among frail older adults, exercise and maintaining self-autonomy are particularly important to reduce fall risk and reduce hospitalizations. It is thought that physical activity that includes strength training to maintain or improve muscle mass throughout aging may reduce muscle loss, an important risk factor for frailty. Supervised exercise is recommended as an effective strategy to treat physical frailty. If physical health is not protected, the quality of life of elderly individuals may decrease along with fragility. It has been observed that people who regularly participate in physical activity in older ages have higher levels of life satisfaction and subjective well-being than those who participate irregularly or intermittently. Yoga is a holistic practice that promotes healing through breathing, movement, strength, flexibility and achieving integrity of spirit, body and mind. Being a meditative practice distinguishes yoga from other typical forms of physical exercise, despite having similar metabolic intensity. Since Yoga aims to create the highest possible state of physical, mental and spiritual health, called Samadhi, many therapeutic processes that balance health occur in the process of achieving this goal. Yoga performed regularly has the potential to improve flexibility, balance and muscle strength in older individuals. It is also known that yoga improves cognitive function in the elderly, helps manage chronic conditions, reduces pain due to osteoarthritis, improves sleep, increases subjective well-being and health-related quality of life. It has been observed that yoga-based practices in the elderly also help maintain breathing and pulse rate, reduce high blood pressure and cortisol levels, and this helps repair stress-related autonomic regulatory reflex mechanisms.

Vinyasa yoga, which is formed by combining breathing flows and exercises with a dance-like flow, is defined in Sanskrit as the art of asanas (postures) related to dynamic meditation of the mind with conscious breathing and body synchronization. It also affects many parameters, affecting a person's health and well-being. The harmony between respiratory mechanics and the musculoskeletal system holistically optimizes body functioning, maintaining serenity and stability as emotional and spiritual calmness of the mind is allowed. In order to maintain the internal balance of the body, in vinyasa yoga, asanas are created as a series of flows in which the breath, described as energy transition called pranayama, is circulated throughout the body. During Vinyasa yoga, breathing continues in its natural flow, but completing the breath at the beginning and end of each asana actually ensures the soft connection between each movement. Depending on the difficulty or depth of physical activity, breathing may deepen or become difficult, but the important and ideal thing is to breathe in a regular rhythm through the nose. This situation, combined with the rhythm of mental and intellectual flows, breathing and asanas, emphasizes the vinyasa aspect of yoga. It is thought that the physical, mental and social effects of fragility can be recycled with a modifiable vinyasa yoga flow for elderly individuals. Despite the increasing prevalence of frailty and its high impact on the elderly, the effects of this condition can be reversed and mitigated with interventions. The American College of Sports Medicine (ACSM) recommends at least 150 minutes per week of moderate-intensity physical activity or 75 minutes per week of vigorous-intensity physical activity for the health benefits of older adults. ACSM recommends moderate to vigorous exercise for cardiovascular health and fitness for healthy adults. In addition, WHO recommends multi-component physical activities that support functional balance and strength exercises at medium or higher intensity, 3 or more days a week, within the weekly physical activities of individuals aged 65 and over, in order to prevent falls and increase functional capacity. Vinyasa yoga has been reported as an alternative moderate-intensity physical activity (50-70% MHR:maximum pulse rate) that meets ACSM criteria and may positively impact cardiovascular health. The metabolic cost of Hatha yoga has been stated to be 2.5 ± 0.8 MET (Metabolic equivalent), corresponding to 49.5 ± 12.2% MHR associated with low-intensity aerobic activity. However, the sequence of sun salutation postures within the typical flow chart of vinyasa yoga has been thought to produce a slightly higher intensity of 2.9 ± 0.77 MET and 54.8 ± 11.8% MHR and may correspond to this when practiced for more than ten minutes . It was also observed that the Hatha yoga practice without Surya Namaskar/sun salutation resulted in approximately 2.07 ± 0.4 MET and 55.98 ± 9.19% MHR, and the sun salutation part corresponded to 3.74 ± 0.70 MET and 66.99 ± 9.99% MHR.

During the healthy aging process, people may need to be guided according to their individual and health characteristics. By supporting this situation with appropriate nursing care, losses can be reduced and optimum health can be maintained. One of the biggest advantages of yoga applied within the scope of nursing care is that the individual's progress is ensured in a controlled manner by preparing a flow in line with appropriate asana selections, taking into account the individual's health condition. Nursing, by its nature, requires a holistic approach to people. Similarly, yoga practice is accepted as a practice that integrates not only physical health but also mind, body and soul.

It is thought that by incorporating the Vinyasa type of yoga, one of the integrative method uses that has just started to participate in the active aging process, into nursing care, it will reduce the exposure of older individuals to risk factors and the positive effects will increase their level of well-being by preventing both multisystemic and multifactorial syndromes. Studies have shown that Vinyasa yoga has a significant effect on transforming negative mood states into positive ones. Physical activity has also been shown to provide mood, emotion and stress reduction benefits.

No studies specifically on vinyasa yoga have been found in the field of nursing. However, when similar holistic practices were examined, Tai-Chi studies were found in the literature for individuals over the age of 60. Yoga, Tai Chi and meditation practices require focus and have been associated with positive changes in brain structure and function, especially in areas related to awareness, attention, executive functions and memory. There are meta-analysis studies showing that Tai-Chi practices have a positive effect on blood pressure by increasing exercise capacity in heart failure patients over the age of 60, and also increase the quality of life by reducing depression.

Since the proposed study has not been found to investigate the effects of vinyasa yoga, which has flows that exercise the musculoskeletal system and also has psychosocial effects, on elderly individuals, it is thought that the data obtained from the research results will contribute to the literature in nursing care by contributing to the active aging process.

ELIGIBILITY:
Inclusion Criteria:

* A student at Ege 3rd Age University
* Those who are between the ages of 65-85,
* Agreeing to participate in the research,
* Open to communication,
* Those with a score of 25 or above according to the mini mental test

Exclusion Criteria:

* Those who are older than 85 and younger than 65,
* Have been meditating regularly in the last year,
* Having attended a 200-hour yoga training program and previously received a certificate,
* Having a chronic disease that will prevent/limit yoga, such as COPD, Asthma, Coronary
* Artery Disease, Heart Failure, and create exercise restrictions.
* Having had a Mini Mental Test within 15 days
* Known history of neoplasia and/or being in the treatment process,
* Having advanced rheumatic or muscular disease

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Groningen Frailty Index | Repeated measurements were made; Groningen Frailty Scale 0.,4.,8. and at the end of the 12. week, it was done 4 times in total.
  "Groningen Frailty Scale" is a scale used to identify frail elderly individuals.The Cronbach's alpha coefficient of the scale was found to be 0.72.GFI is a 15-item screening tool that measures physical, cognitive, psychosocial and polypharmacy frailty in the form of professional and self-report to determine the level of frailty. Eight items have two response categories (yes / no), six items have three response categories (yes / sometimes / no), and one item has a Likert type response category (1-10). A high GFI total score indicates a high level of frailty. The total score obtained from the scale varies between 0 and 15, and higher scores indicate more fragility. The answer to each item has 0 or 1 point; 1 indicates a problem with vulnerability and fondness.
Skeletal muscle and appendicular muscle mass measurement from anthropometric (physiological parameter) measurements with Bioelectrical Impedance Analysis | These measurements were applied as pretest and posttest. It was applied at week 0 and week 12.
  It is the measurement of tissues in the body, such as muscle and fat, which are rich in liquid electrolytes, with a portable device. Although there is no direct tissue measurement, accurate results can be achieved within the framework of certain standards that affect the conductivity state.With BIA measurements, skeletal muscle mass (Skeletal Muscle Mass = SMM), appendicular muscle mass (Apendicular skeletal muscle mass = ASM) and the indices SMI and ASMI, which are formed by dividing the square meter of these measurements to the height, can be measured. ASM is 15 kg and above in a healthy adult woman; For men, it should be 20 kg and above. For ASMI, 7 kg/m2 and above in men and 5.5 kg/m2 and above in women are considered normal values. Both low muscle strength and low muscle mass suggest a diagnosis of sarcopenia in individuals.
Hand Grip Test | These measurements were applied as pretest and posttest. It was applied at week 0 and week 12.
  The isokinetic dynamometer measurement test, which is considered the gold standard in the evaluation of muscle strength, is performed by examining the highest force realized with the flexion of all hands and fingers under biokinetic conditions.
4-Meter Walk Gait Speed Test | These measurements were applied as pretest and posttest. It was applied at week 0 and week 12.
  In the 4 meter walking test; The individual is expected to walk a distance of 4 meters in less than 5 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Adaiçi, PhD Student, Principal Investigator — Ege University; Nazmiye Çıray, Asst. Prof., Study Director — Ege University; Fisun Şenzun Aykar, Prof., Study Director — Izmir Tinaztepe University
Locations (1):
- Ege University, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Since it is a doctoral thesis study, it will be shared at the Turkish Higher Education Institution National Thesis Center when the thesis process is completed.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: It can be used in accordance with the time it was published in the Turkish National Thesis Center (YÖKTEZ).
Access Criteria: It is available as of the time it is published in the Turkish National Thesis Center (YÖKTEZ).
URL: https://tez.yok.gov.tr/UlusalTezMerkezi/

REFERENCES:
- [Result] Lau C, Yu R, Woo J. Effects of a 12-Week Hatha Yoga Intervention on Metabolic Risk and Quality of Life in Hong Kong Chinese Adults with and without Metabolic Syndrome. PLoS One. 2015 Jun 25;10(6):e0130731. doi: 10.1371/journal.pone.0130731. eCollection 2015. PMID 26111165
- [Result] DiBenedetto M, Innes KE, Taylor AG, Rodeheaver PF, Boxer JA, Wright HJ, Kerrigan DC. Effect of a gentle Iyengar yoga program on gait in the elderly: an exploratory study. Arch Phys Med Rehabil. 2005 Sep;86(9):1830-7. doi: 10.1016/j.apmr.2005.03.011. PMID 16181950
- [Result] Ni M, Mooney K, Richards L, Balachandran A, Sun M, Harriell K, Potiaumpai M, Signorile JF. Comparative impacts of Tai Chi, balance training, and a specially-designed yoga program on balance in older fallers. Arch Phys Med Rehabil. 2014 Sep;95(9):1620-1628.e30. doi: 10.1016/j.apmr.2014.04.022. Epub 2014 May 14. PMID 24835753
- [Result] Pina AA, Shadiow J, Tobi Fadeyi A, Chavez A, Hunter SD. The acute effects of vinyasa flow yoga on vascular function, lipid and glucose concentrations, and mood. Complement Ther Med. 2021 Jan;56:102585. doi: 10.1016/j.ctim.2020.102585. Epub 2020 Oct 7. PMID 33197660
- [Result] Miller SM, Hui-Lio C, Taylor-Piliae RE. Health Benefits of Tai Chi Exercise: A Guide for Nurses. Nurs Clin North Am. 2020 Dec;55(4):581-600. doi: 10.1016/j.cnur.2020.07.002. Epub 2020 Oct 13. PMID 33131634
- [Result] Shin S. Meta-Analysis of the Effect of Yoga Practice on Physical Fitness in the Elderly. Int J Environ Res Public Health. 2021 Nov 6;18(21):11663. doi: 10.3390/ijerph182111663. PMID 34770176